CLINICAL TRIAL: NCT01038245
Title: Quantitation of Human Cerebral Nicotinie Receptors With 2[18F]FA-85380 and PET Healthy Non-smokers and Ex-Smokers and in Heavy and Light Situational Smokers
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903383; 03-DA-N383
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-11-18

CONDITIONS: Nicotine Addiction
Keywords: Receptor Up-Regulation; Smoking; Nicotine; Neuroimaging
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

SUMMARY:
Background:

- Central nicotinic acetylcholine receptors (nAChRs) are primary targets for the action of nicotine. In addition to being involved in tobacco dependence, they are also involved in a variety of brain disorders, including Alzheimer's and Parkinson's diseases. Researchers are interested in developing better ways to study the action of nAChRs to improve treatments for smoking cessation and other problems affected by these receptors. These new study methods may involve different approaches to positron emission tomography (PET) scanning, which can show brain activity related to nAChRs.

Objectives:

- To evaluate appropriate and useful doses of radiotracers used in PET scanning of nAChRs in the brains of nonsmokers/former smokers, light smokers, and heavy smokers.

Eligibility:

- Individuals between 18 and 50 years of age who fall into one of the following groups: (1) nonsmokers or former smokers who have not smoked for the past 2 years, (2) light/situational smokers, or (3) heavy smokers (at least 15 cigarettes/day for the past 2 years).

Design:

* Each participant will undergo up to three PET studies, given approximately1 month apart. Each study will take approximately 8 hours to complete.
* Participants will provide urine and breath samples before the study and at the start of the study, which will be tested for chemicals that may interfere with the study.
* Depending on the study, some of the smoking participants may receive a nicotine patch to wear during the PET scan.
* On the day of the study, participants will receive a dose of a radiotracer (a drug used in PET scanning) given either as a single injection or as an injection followed by a continuous infusion, and will have a series of PET scans over the next 7 hours and provide blood samples during that time.
* Participants will return for a follow-up visit 1 month after the end of the study.

DETAILED DESCRIPTION:
Background: Central nicotinic acetylcholine receptors (nAChRs) mediate a variety of brain functions and have been implicated in the pathophysiology of Alzheimer's and Parkinson's diseases, other CNS disorders (Tourette's syndrome, epilepsy, etc.), and nicotine dependence. These receptors are the primary target for the action of nicotine, which is believed to cause tobacco dependence. The ability to quantitatively image nAChRs with PET in humans would allow scientists to monitor the nAChRs in vivo during nicotine dependence and smoking cessation and to determine the receptor occupancy by nicotine for different types of nicotine replacement therapy (NRT). Recently completed studies demonstrated the feasibility of imaging nAChRs in the human brain with 2[18F]FA-85380 and showed that each participant could receive up to 4 injections of 5 mCi/70 kg without exceeding dosimetry limits imposed by the FDA and the NIH Radiation Safety Committee.

Scientific Goal: The aims of the proposed study are 1) to compare the total volumes of distribution for 2[18F]FA-85380 and volumes of distribution for specific binding compartment (an estimate of nAChR densities) in brains of light and heavy smokers and 2) to develop a simplified PET procedure that is more comfortable for the human participants and that maintains the ability to accurately quantify nAChR binding in vivo.

Study Population: Healthy adult participants (non-smokers or exsmokers and light (situational) and heavy smokers), males and females between 18 and 50 years of age, will be recruited for this study. The goal is to complete studies of 12 controls (non-smokers or exsmokers), 12 light smokers and 12 heavy smokers.

Experimental Design and Method: After being medically cleared and giving informed consent, each participant will undergo up to three PET studies. In each study, the participant will receive a 5 mCi/70 kg dose of the radioligand, 2[18F]FA-85380-Injection. For one of the studies, the participants who smoke will receive nicotine by a nicotine patch (Nicoderm), applied approximately 4 h before the scan. The patch will be removed 12 h after it is applied. For two studies (one without and one with nicotine), participants who smoke will receive the radioligand as a bolus injection. Six of the participants who do not currently smoke (control group) will receive the radioligand as a bolus injection twice without nicotine either time. For the third study, all participants will receive the radioligand as a bolus injection followed by a continuous infusion (bolus injection/infusion combination). Six of the participants who do not currently smoke (control group) will receive the radioligand as a bolus plus infusion injection twice. For each study, a series of brain PET scans will be acquired for 8 h beginning at the time of the injection. The data from the PET scans without and with nicotine patch (smokers only) will be used to determine the total and non-specific accumulation of radioactivity in the brain. The data from the equivalent two PET scans for the controls will be used to determine the test-retest reliability of the measure. The data from the PET scans acquired from the bolus/infusion paradigm will be used to demonstrate the feasibility of a shorter scanning period for quantitation studies. It is anticipated that several of the participants will choose not to continue after the first scan. The study design accommodates this expectation.

Benefits to participants and/or society: This protocol will provide no direct benefits to the research participants other than routine medical screening and attention from the research staff. The knowledge gained in this study may lead to the availability of an agent for external monitoring of nAChRs using PET. This agent would be a valuable tool for determining the dynamics of nAChRs in nicotine dependence and smoking cessation.

Risks to participants: There are risks related to the PET scans in general, involving exposure to radiation, arterial catheterization and venous catheterization. In addition, there are risks related to the administration of this radiopharmaceutical and from exposure to nicotine. Medical supervision will be provided throughout the study. A plan for monitoring potential side effects of this radiotracer is given.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: Subjects will be male and female volunteers aged 18 to 50 years.
* All subjects must have a stable point of contact and must agree to participate in three PET studies at approximately 4-week intervals.
* All participants in the light or heavy smoker groups must have smoking experience. Those in the heavy smoker group must smoke at least 15 cigarettes/day and have smoked for at least the last 2 consecutive years. Those participants in the light smoker group should be situational smokers (those who often smoke while consuming alcohol or in another type of situation, but who do not smoke daily). Light smokers should have not smoked more than 1 cigarette in the week before starting the medical screening process and agree to not smoke for the week before the first PET study (except for the single cigarette we ask them to smoke). Participants in the heavy smoker group should have experience with abstaining from smoking for at least 48 h. Subjects in the control group must be nonsmokers or have ceased smoking at least two years before the start of the study.

EXCLUSION CRITERIA:

* Weight: Anyone weighing more than 300 lbs is excluded from the study.
* Psychiatric disease: DSM-IV criteria will be used (American Psychiatric Association, 1994). No subject with a current axis I diagnosis will be allowed. No subject with known claustrophobia will be allowed.
* History of Drug Abuse: Volunteers reporting current or having a significant history of illicit drug abuse (single illicit substance use of more than 30 times in a lifetime for any given substance, except marijuana) will be excluded from the study. However, if the use was greater than 10 times in a lifetime, it must have occurred more than 10 years before enrollment in this protocol. Subjects may use moderate amounts of alcohol and caffeine and smoke an occasional marijuana cigarette. Moderate alcohol use will be defined as less than fourteen drinks of liquor (1.5 oz) or the equivalent beer (12 oz) or wine (5 oz) per week. Moderate caffeine use will be defined as less than 500 mg of caffeine per day, where 100 mg is equivalent to 1 serving of coffee (5 oz serving), 2.5 servings (12 oz serving) of caffeinated soft drinks, or 2.5 servings of tea (5 oz serving). Occasional marijuana use will be defined as less than or equal to two marijuana cigarettes/month.
* Current Medication Use: Volunteers may not currently use chronic (daily or for more than 10/14 days in the last month) prescription or over the counter medications, (including, but not limited to, anti-hypertensive, anti-allergy, pain).
* CNS disease: History of known structural brain abnormalities (e.g., neoplasm, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), history of head trauma (defined as documented loss of consciousness > 5 min or injury requiring hospitalization), history of seizures as an adult, sleep apnea.
* Cardiovascular, pulmonary, or systemic disease: Repeated (measured on three separate occasions) diastolic blood pressure > 90 mm Hg, or systolic blood pressure > 150 mm Hg, known arrhythmia, symptomatic or known coronary artery disease; history of endocarditis, cerebral embolism, obstructive pulmonary disease, asthma, active tuberculosis, known endocrine disease (derangements in adrenal, thyroid, bone or reproductive function) known chronic renal or hepatic dysfunction, known HIV seropositive, known current autoimmune disease involving the CNS, type I diabetes mellitus, current gastrointestinal disease, gastritis or ulcers.
* Special considerations for female subjects. Female participants who are currently pregnant or nursing will not be allowed to participate in this study because of potential damage to the fetus or baby from the radiation. Female subjects will be given a serum pregnancy test (quantitative beta HCG) within 24 hours of each PET study.
* Radiation exposure: Any subject who has participated in any research studies in which he/she received a radiation exposure that would result in combination with the present study, in a total effective radiation exposure (from research studies) exceeding 3.0 rem in a 13-week period or 5.0 rem in a year.
* Lack of bilateral arterial patency: Evidence of inadequate patency of radial and lunar arteries, determined by either Doppler flow measurements or a positive Allen's test, is an exclusionary criterion for insertion of an arterial catheter.
* Women who are pregnant or lactating and children under the age of 18 will be excluded to avoid unnecessary exposure to radiation to these populations.
* Presence in body of metallic implants or materials that could be moved by the magnet of the MRI scanner: pacemakers, surgical implants, aneurysm clips, dental braces, bullet(s) or other metallic materials.
* Miscellaneous exclusionary criteria: Body mass index less than 19 or greater than 30. Hematocrit < 39.0 for males or < 36.0 for females.
* Novocain allergy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2003-07-08; Study Completion 2011-11-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States